CLINICAL TRIAL: NCT02910440
Title: A Randomized, Investigator-blinded, Non-inferiority, Multicenter Study Evaluating the Safety and Efficacy of DCL-101 Compared to GoLYTELY in Adult Outpatients Undergoing Routine Colonoscopy
Brief Title: A Safety and Efficacy Study of DCL-101 Compared to GoLYTELY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dark Canyon Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCL-101-201
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Bowel Preparation Before Colonoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator

ARMS (2):
- DCL-101 (Experimental)
  Interventions: Drug: DCL-101 vs Golytely
- GoLytely (Active Comparator)
  Interventions: Drug: DCL-101 vs Golytely

INTERVENTIONS:
Drug: DCL-101 vs Golytely

SUMMARY:
The primary objective of this Phase 2 Study was to compare the safety of 3 liter(L) and 4 liter(L) split dose DCL-101 to split dose 4L GoLYTELY in patients preparing for colonoscopy, with secondary objectives to assess tolerability and bowel cleansing efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating females, 18 to 75 years of age. Females of child bearing potential must have a negative urine pregnancy test prior to randomization, and must use a hormonal (oral, implantable or injectable) or barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
2. Routine, non-urgent, screening or surveillance colonoscopy is indicated and scheduled.
3. Ability of subject to participate fully in all aspects of this clinical trial, including ability and willingness to swallow capsules.
4. Informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization will be obtained and documented from all subjects prior to the start of any study-specific procedures.

Exclusion Criteria:

1. Known hypersensitivity or allergy to any of the components of GoLYTELY or DCL-101
2. Actual or suspected ileus, gastrointestinal obstruction or other major structural gastrointestinal disorders, esophageal stricture, gastric retention, bowel perforation, toxic colitis, ischemic colitis, infectious colitis, toxic mega-colon, or inflammatory bowel disease. Diverticulitis within the past 6 weeks
3. Current or former tobacco users
4. Prior colorectal surgery, esophageal surgery, or gastric surgery. This includes colectomy in the past, colostomy, ulcer surgery (antrectomy or pyloroplasty) or bariatric surgery, including lap band or fundoplication
5. Chronic constipation, gastroparesis, esophageal motility disorders or other gut dysmotility disorders
6. Requiring medications that cannot have the administration schedule safely altered to be compatible with bowel preparation
7. Current or history within the past year of any ongoing clinically relevant electrocardiogram abnormalities
8. Clinically significant electrolyte abnormalities during Screening, defined by the range of normal of the central laboratory
9. Significant psychiatric illness
10. Renal failure or chronic kidney disease (creatinine clearance less than 50 mL/min, unstable angina, acute coronary syndrome/congestive heart failure (New York Heart Association Functional Classification grade III or IV), ascites
11. Received any investigational therapy within 60 days of randomization
12. Blood donation within 56 days prior to randomization
13. Plasma donation within 7 days prior to randomization
14. Received luminal contrast agents such as barium or water-soluble oral contrast agent within 21 days prior to randomization
15. Known to have an impaired gag reflex, or prone to regurgitation or aspiration
16. Serious underlying disease that in the opinion of the investigator may interfere with the subject's ability to participate fully in the study
17. History of alcohol or drug abuse that in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures
18. Pregnant or lactating women
19. Prior enrolment in the current study and had received study treatment
20. Cognitive barriers that in the opinion of the investigator may interfere with the subject's ability to participate fully in the study
21. Inability to either read or understand English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Graded Adverse Events | 2-6 hours after completion of investigational agent administration
  Scale: Common Terminology Criteria for Adverse Events, a 5-point scale with Grade 1 equal to "mild" and Grade 5 equal to "death"

SECONDARY OUTCOMES:
Incidence of Graded Adverse Events | 1-2 days after completion of investigational agent administration
  Scale: Common Terminology Criteria for Adverse Events, a 5-point scale with Grade 1 equal to "mild" and Grade 5 equal to "death"
Incidence of Graded Adverse Events | 7 days after completion of investigational agent administration
  Scale: Common Terminology Criteria for Adverse Events, a 5-point scale with Grade 1 equal to "mild" and Grade 5 equal to "death"
Incidence of Serious Adverse Events | 2-6 hours after completion of investigational agent administration
  Scale: Events that are life-threatening, lead to hospitalization, cause permanent injury, or death
Incidence of Serious Adverse Events | 1-2 days after completion of investigational agent administration
  Scale: Events that are life-threatening, lead to hospitalization, cause permanent injury, or death
Incidence of Serious Adverse Events | 7 days after completion of investigational agent administration
  Scale: Events that are life-threatening, lead to hospitalization, cause permanent injury, or death
Incidence of abnormal blood chemistries | 2-6 hours after completion of investigational agent administration
  Scale: Normal range, as established by study reference laboratory
Incidence of abnormal blood chemistries | 1-2 days after completion of investigational agent administration
  Scale: Normal range, as established by study reference laboratory
Incidence of abnormal blood chemistries | 7 days after completion of investigational agent administration
  Scale: Normal range, as established by study reference laboratory
Incidence of abnormal urinalysis | 2-6 hours after completion of investigational agent administration
  Scale: Normal range, as established by study reference laboratory
Incidence of abnormal urinalysis | 1-2 days after completion of investigational agent administration
  Scale: Normal range, as established by study reference laboratory
Incidence of abnormal urinalysis | 7 days after completion of investigational agent administration
  Scale: Normal range, as established by study reference laboratory
Incidence of clinically significant electrocardiogram (ECG) changes | 2-6 hours after completion of investigational agent administration
  Scale: Comparison with baseline ECG
Incidence of clinically significant electrocardiogram (ECG) changes | 7 days after completion of investigational agent administration
  Scale: Comparison with baseline ECG
Incidence of orthostatic hypotension | 2-6 hours after completion of investigational agent administration
  Scale: Defined as a drop of >20 mmHg of the systolic blood pressure, or a drop of > 10 mm Hg of the diastolic blood pressure, when going from a supine position to standing for 2 minutes, and measured standing.
Incidence of orthostatic hypotension | 1-2 days after completion of investigational agent administration
  Scale: Defined as a drop of >20 mmHg of the systolic blood pressure, or a drop of > 10 mm Hg of the diastolic blood pressure, when going from a supine position to standing for 2 minutes, and measured standing.
Incidence of orthostatic hypotension | 7 days after completion of investigational agent administration
  Scale: Defined as a drop of >20 mmHg of the systolic blood pressure, or a drop of > 10 mm Hg of the diastolic blood pressure, when going from a supine position to standing for 2 minutes, and measured standing.
Between group difference in the aggregate tolerability score (ATS) of the Lawrance Colonoscopy Preparation Patient Tolerability Questionnaire | 2-6 hours after completion of investigational agent administration
  The Bowel-Preparation Tolerability Questionnaire by Lawrance et. al. (Lawrance Instrument) is a validated questionnaire asking patients to score nine symptoms during bowel preparation on a 5-point Likert scale. These symptom scores are summed for all nine symptoms to arrive at an aggregate tolerability score (ATS), with a lower ATS indicating better tolerability.
Between group difference in score in individual aspects of the Lawrance Colonoscopy Preparation Patient Tolerability Questionnaire | 2-6 hours after completion of investigational agent administration
  Nine symptoms during bowel preparation on a 5-point Likert scale by patient
Between group difference in the Symptom Score of the Mayo Clinic Bowel Prep Tolerability Questionnaire | 2-6 hours after completion of investigational agent administration
  The Mayo Clinic Bowel Prep Tolerability Questionnaire (Mayo Instrument) is a validated questionnaire containing 8 items including questions addressing tolerability, ability to consume the entire dose, and willingness to use again. Patients are also asked to score seven symptoms during bowel preparation on a 4-point Likert scale, which are averaged to determine a Symptom Score.
Proportion of subjects compliant with 90% of the study treatment regimen | At time of colonoscopy
  Consumption of a minimum of 90% of GoLYTELY solution or 90% of DCL-101 kit, as applicable
Proportion of subjects compliant with 100% of the study treatment regimen | At time of colonoscopy
  Consumption of 100% of GoLYTELY solution or 100% of DCL-101 kit, as applicable.
The mean total score on the centrally read Ottawa Bowel Preparation Quality Scale (OBPQS) | At time of colonoscopy
The proportion of subjects achieving an OBPQS score of 2 or less (excellent), with no segment score greater than 1, on the centrally read OBPQS | At time of colonoscopy
The mean segmental scores and the mean colonic fluid quantity score from the centrally read OBPQS | At time of colonoscopy
The proportion of subjects achieving a score of 8 or greater on the Boston Bowel Preparation Scale (BBPS) | At time of colonoscopy
The proportion of subjects with segmental scores of 2 or greater on the BBPS for every one of the segments | At time of colonoscopy
The mean total score on the BBPS | At time of colonoscopy
The Aronchick score (excellent, good, fair, poor, unsatisfactory) | At time of colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Philip N Calvillo, Study Chair — Alimentiv Inc.
Locations (5):
- United States (5):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Asheville Gastroenterology, Asheville, North Carolina
  - Cumberland Research Associates LLC, Fayetteville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Trial Management Associates, Wilmington, North Carolina

REFERENCES:
- [Derived] Bachwich DR, Lewis JD, Kowal VO, Jacobson BC, Calderwood AH, Kochman ML. A Phase 2 Randomized Trial of DCL-101, a Novel Pill-Based Colonoscopy Prep, vs 4L Polyethylene Glycol-Electrolyte Solution. Clin Transl Gastroenterol. 2020 Dec;11(12):e00264. doi: 10.14309/ctg.0000000000000264. PMID 33512795